CLINICAL TRIAL: NCT02391935
Title: Randomized, Double-blind, Placebo-controlled, Single-centre, Phase I Safety Study of Intradermal Injections of RCS-01 in Male and Female Subjects (50 to 65 Years Old)
Brief Title: Study of Intradermal Injections of RCS-01 in Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RepliCel Life Sciences, Inc. (Industry)
Collaborators: JensonR+ Limited (Unknown); PHARMALOG Institut für klinische Forschung GmbH (Unknown); Syreon Corporation (Industry); Innovacell Biotechnologie AG (Industry); Datinf GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RCS-01-001-2014
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Intrinsic Aging of Skin; Skin Wrinkling; Solar Degeneration of Skin
Keywords: Chronic Effect of Ultraviolet Radiation on Normal Skin (Photo-aging)

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RCS-01 (Experimental): Cultured, autologous hair follicle cells suspended in cryomedium
  Interventions: Drug: RCS-01; Drug: Placebo; Device: Sham injection
- Placebo (Placebo Comparator): cryomedium
  Interventions: Drug: Placebo; Device: Sham injection

INTERVENTIONS:
Drug: RCS-01 — Cultured, autologous hair follicle cells suspended in cryomedium
  Arms: RCS-01
Drug: Placebo — Cryomedium
Device: Sham injection — skin penetration of the needle without injection of liquid

SUMMARY:
The primary purpose of this study is to assess the safety profile of RCS-01 injections as compared to placebo injections. This study will also measure the impact these injections will have on skin markers related to aging through evaluation of gene expression profiles.

30 participants will be selected for this study based on their health status, current/past medications, and ability to adhere to protocol-related requirements. At the first visit and after providing informed consent, participants are evaluated against the study inclusion/exclusion criteria and provide blood samples for screening assessments (including virology). If suitable for study participation, participants will provide a biopsy from the scalp from which RCS-01 will be prepared and will have four treatment evaluation sites identified on their buttocks, two on each side.

Study participants will be randomized to one of two treatment subgroups. Participants in the RCS-01 Subgroup (n=24) will receive injections of RCS-01 or placebo or a 'sham' injection (a needle penetration without injection of liquid). Participants in the the Placebo Subgroup (n= 6) will be randomized to receive only injections of placebo or sham injections.

Baseline evaluations of subjects' overall health and skin condition at treatment sites on their buttocks will be performed before receipt of injections at Day 0. In addition to injections delivered at Day 0, the pre-selected treatment evaluation sites will receive intradermal injections of RCS-01 or placebo (cryomedium) or a sham injection four (4) and eight (8) weeks after Day 0 according to a randomization schedule for a total of three (3) injections per treatment site.

All participants will return to the clinic for at least 9 visits during the 52-week follow-up period to monitor long-term safety. At the 12-week time point, 18 randomly-selected participants from the RCS-01 Subgroup will provide biopsies from all injection sites for analysis of skin markers related to aging. At the 26-week time point, the remaining participants will provide biopsies of all injection sites for histopathological analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female Caucasian in good health between the age of 50 and 65 years.
2. Female subjects must be post-menopausal for at least one year or surgically sterile.
3. Signed and dated informed consent and willingness to attend all study visits and complete all procedures required by this protocol.
4. The treatment evaluation sites are of uniform skin color without erythema, dark pigmentation or scars that may confound study results.

Exclusion Criteria:

1. Any transient skin disorder or infections (e.g. pyoderma, tinea corporis, contact or irritative dermatitis, scleroderma etc.) within 20 cm of the treatment evaluation sites or the presence of tattoos near the treatment sites.
2. Subjects diagnosed with psoriasis, lichen planus, vitiligo, systemic scleroderma, or lupus erythematosus.
3. Any condition that, in the investigator's opinion, would impact subject's safety and/or a subject's ability to complete all study related procedures.
4. History of infection with or positive serology results for human immunodeficiency virus (HIV), hepatitis B or C, or syphilis.
5. Presence/history of hypertrophic scars and/or keloids.
6. Subjects diagnosed with cancer with or without chemotherapy treatment within 3 years prior enrollment.
7. Women who are pregnant or nursing.
8. Current use of any medications not permitted in the study
9. Ongoing or recent participation in a cosmetic and/or clinical research study prior to enrolment.
10. Subject not agreeing to avoid UV exposure (sun, solarium) on the nude buttocks during the study period.
11. Known allergy or hypersensitivity to human serum albumin, DMSO, gentamicin, material of bovine origin and/or local anesthetics.
12. Close affiliation with the investigational site (e.g., a close relative of the investigator or a possibly dependent person (e.g., employee or student of the investigational site)).
13. Subjects diagnosed with coagulopathies or significant thrombocytopenia

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-10-10 (Actual); Primary Completion 2017-07-12 (Actual); Study Completion 2017-07-12 (Actual)

PRIMARY OUTCOMES:
Incidence of local adverse events | 52 weeks after first injection
  Within-patient comparison of the local (reported at treatment evaluation sites) adverse event profile between treatment evaluation sites treated with RCS-01 or placebo. The local adverse event profile is defined by the incidence, relationship to treatment, severity and seriousness of adverse events reported at the treatment evaluation sites.

SECONDARY OUTCOMES:
Incidence of adverse events | 52 weeks after first injection
  Between-subject comparison of the systemic (not reported at treatment evaluation sites) adverse event profile between participants in the RCS-01 Subgroup versus Placebo Subgroup.
Incidence of abnormalities in skin structure | 52 weeks after first injection
  A within-patient and between patient comparison of histology results from analyses performed on biopsies obtained from treatment evaluation sites.
Incidence of changes in markers related to skin aging | 12 weeks after first injection
  Markers to be assessed include fibrillar collagen type I (COL 1A1, COL 1A2) and type III (COL 3A1), transforming growth factor beta1, connective tissue growth factor, matrix metalloproteinases 1, 3 and 9, tissue inhibitor of matrix metalloproteinase 1 and lumican . Incidence of changes within- and between-participants.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Marini, MD, Principal Investigator — IUF Leibniz-Institut für umweltmedizinische Forschung gGmbH
Locations (1):
- IUF Leibniz-Institut für umweltmedizinische Forschung gGmbH, Düsseldorf, Germany

REFERENCES:
- See also: RepliCel Life Sciences, Inc. Website — http://www.replicel.com